CLINICAL TRIAL: NCT05772728
Title: A Multicenter, Single-arm, Open Clinical Efficacy Observational Study of Cidapenem Combined With Azacitidine and Mitoxantrone Liposome (CAM) Regimen for Relapsed/Refractory Intra-nodal Follicular Adjuvant T-cell Lymphoma (nTFHL)
Brief Title: Chidamide Combined With Azacitidine and Mitoxantrone Liposome in the Treatment of Relapsed/Refractory (nTFHL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-571
Record Dates: First submitted 2022-12-29; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Azacitidine; Clinical Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAG Group (Experimental): Cidapenem combined with azacitidine and mitoxantrone liposomes
  Interventions: Drug: Cidapenem combined with azacitidine and mitoxantrone liposome (CAM) regimen

INTERVENTIONS:
Drug: Cidapenem combined with azacitidine and mitoxantrone liposome (CAM) regimen — CAM regimen (every 21 days as a treatment cycle). Cetapenem 20 mg orally twice weekly Azacitidine 75 mg/m2 subcutaneously d1-7 Mitoxantrone liposomes 20 mg/m2 intravenous d6
  Other Names: CAM

SUMMARY:
Intranodal follicular adjuvant T-cell lymphoma (nTFHL) is a type of peripheral T-cell lymphoma (PTCL) that is a new subtype in WHO 2022, which includes 3 categories corresponding to previous angioimmunoblast T-cell lymphoma (AITL), follicular T-cell lymphoma, and PTCL with TFH phenotype, named nTFHL-angioblast type ( nTFHL-AI), nTFHL-follicular (nTFHL-F), and nTFHL-non-specific (nTFH-NOS), respectively.1 nTFHL-AI has a relatively high incidence in PTCL, accounting for about 25-30% of cases, with an aggressive clinical presentation, often with multisystem involvement and with immune system abnormalities. nTFHL shares common immunophenotypic features, namely TFH cell phenotype: CD279/PD1, CD10, BCL6, CXCL13, ICOS, SAP, and CCR5, and at least 2 of the stated immune markers combined with CD4 positivity are required for the diagnosis of nTFHL.1, TFH cell and nTFHL cell also share similar reproducible genetic abnormalities, such as RHOA G17V, DNMT3A, IDH2, TET2, often involving epigenetic genetic abnormalities 2, especially abnormalities of DNMT3A, IDH2, and TET2 are more frequent in myeloid disorders.

Basic studies have shown that cidabenamide and anthracyclines have synergistic effects to promote apoptosis in PTCL cells; and the adverse events of the two do not completely overlap, suggesting that a mitoxantrone liposome-based regimen combined with cidabenamide for PTCL may have a better clinical benefit.

Based on the above findings, the investigators propose to further investigate the efficacy and safety of cidapenem combined with azacitidine and mitoxantrone liposome (CAM) regimen, i.e., cidapenem combined with azacitidine dual epigenetic modulation on the basis of mitoxantrone liposome, in the treatment of patients with R/R nTFHL using a randomized, prospective, multicenter phase II clinical trial, which is expected to further improve ORR, PFS and OS.

DETAILED DESCRIPTION:
Induction treatment period. Cetapenem 20 mg orally twice a week Azacitidine 75 mg/m2 subcutaneously d1-7 Mitoxantrone liposomes 20 mg/m2 intravenous d6

1 treatment cycle every 21 days. Maintenance treatment period: cidabendiamide 20 mg orally twice weekly/28 days Cycle

ELIGIBILITY:
Inclusion Criteria:

1. R/R nTFHL confirmed by pathological tissue, with diagnostic criteria referring to the 2022 WHO diagnostic criteria.
2. Patients who have undergone at least one previous systemic treatment (including chemotherapy, HSCT, etc.) without remission or relapse after remission.
3. Signed written informed consent and who are able to comply with the visits and related procedures specified in the protocol.
4. whole-body PET/CT performed 28 days prior to study entry, which must have at least 1 evaluable or measurable lesion meeting Lugano 2014 criteria: lymph node lesions, measurable lymph nodes need to be >1.5 cm in length; non-lymphoid lesions, measurable extra-nodal lesions need to be >1.0 cm in length.
5. with a PS score of 0 to 2 according to ECOG
6. with adequate organ and bone marrow function, defined as follows: neutrophil count ≥ 1.5×109/L, platelet count ≥ 75×109/L, and hemoglobin ≥ 80 g/L (relaxed to ≥ 1.0×109/L for neutrophil count, ≥ 50×109/L for platelet count, and ≥ 75 g/L for hemoglobin in patients with bone marrow involvement);
7. Liver and kidney function: serum creatinine (Cr) ≤ 1.5 times the upper limit of normal value; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal value (≤ 5 times the upper limit of normal value for patients with liver invasion); total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver invasion);
8. life expectancy of more than 3 months
9. age 18 to 75 years.

Exclusion Criteria:

1. Subjects with a history of prior antitumor therapy that is one of the following.

   1. Previous recipients of mitoxantrone or mitoxantrone liposomes.
   2. Prior treatment with doxorubicin or other anthracyclines with a total cumulative dose of doxorubicin > 360 mg/m2 (other anthracyclines converted to 1 mg doxorubicin equivalent to 2 mg epirubicin).
   3. Patients who have received autologous hematopoietic stem cell transplantation (ASCT) within 100 days of the first dose, or who have received allogeneic hematopoietic stem cell transplantation.
   4. have received antitumor therapy (including chemotherapy, targeted therapy, hormonal therapy, administration of herbal medicine with antitumor activity, etc.) or participated in other clinical trials and received clinical trial medication within 4 weeks prior to the first administration of this study drug.
2. Hypersensitivity reaction to any investigational drug or its components.
3. Uncontrollable systemic disease (e.g., progressive infection, uncontrollable hypertension, diabetes mellitus, etc.).
4. Cardiac function and disease consistent with one of the following.

   1. Long QTc syndrome or QTc interval >480 ms.
   2. Complete left bundle branch block, second or third degree atrioventricular block.
   3. Severe, uncontrolled arrhythmias requiring drug therapy.
   4. American New York Heart Association classification ≥ Class III.
   5. Cardiac ejection fraction (LVEF) less than 50%.
   6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia, or any other arrhythmia requiring treatment, history of clinically severe pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities within 6 months prior to recruitment.
5. Active hepatitis B and C infection (positive hepatitis B virus surface antigen and hepatitis B virus DNA greater than 1 x 103 copies/mL; hepatitis C virus RNA greater than 1 x 103 copies/mL).
6. Human immunodeficiency virus (HIV) infection (HIV antibody positive).
7. previous or current concurrent other malignancies (in addition to effectively controlled non-melanoma basal cell carcinoma of the skin, breast/cervical carcinoma in situ and other malignancies that have not been treated and also effectively controlled within the last five years)
8. Primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment.
9. Pregnant and lactating women and patients of childbearing age who do not wish to use contraception
10. Persons with mental disorders/unable to obtain informed consent.
11. Those who are judged by the investigator to be unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective Response Rate

SECONDARY OUTCOMES:
2 year PFS rate | 2 years
  2 year PFS rate
2 year OS rate | 2 years
  2 year OS rate
DOR | 2 years
  Duration of remission